CLINICAL TRIAL: NCT06988618
Title: Real-world Experience on Using Nemolizumab in the Treatment of Moderate-to- Severe Prurigo Nodularis in Adults
Acronym: RE-UNITE PN
Status: Recruiting | Type: Observational
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: SPR207807
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Prurigo Nodularis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nemolizumab: Participants with moderate-to-severe PN who are receiving nemolizumab (Nemluvio®) in routine clinical practice will be observed for approximately 12 months.

SUMMARY:
The main aim of this study is to assess real-world effectiveness of nemolizumab in Prurigo nodularis (PN) as measured by investigator and patient reported outcome (PRO) in clinical practice at Month 6.

DETAILED DESCRIPTION:
This prospective, multicenter, non-interventional study (NIS) seeks to evaluate PN treatment with nemolizumab (Nemluvio®) in adults over an approximately 12 month period using physician assessments in routine clinical practice and PRO measures. Treatment with nemolizumab will be determined solely by the participant's physician prior to study enrollment. No additional visits, procedures, or laboratory tests are required outside of routine clinical practice.

The visit structure is not defined by the study protocol but is determined by routine medical practice. The visit schedule is intended to facilitate a systematic data assessment according to clinical routine. A sub-study will be completed in Germany and the UK at selected sites in which participants will complete the Peak pruritus (PP) numerical rating scale (NRS) and Sleep Disturbance (SD) NRS on a daily basis from Day -1 to Day 14. Data collection will occur remotely and no clinic visits will be required.

ELIGIBILITY:
Inclusion Criteria:

* Participants who, according to the treating physician's decision and in line with the local package label, are newly initiated on nemolizumab (Nemluvio®) for the treatment of PN.
* Participants greater than or equal to (>=) 18 years of age.
* Participants who signed the written informed consent form (ICF).

Exclusion Criteria:

* Have contraindication(s) for the use of nemolizumab (Nemluvio®) according to the local package label;
* Participants who received treatment with a drug under clinical development/ investigation within 3 months prior to baseline.
* Participants who received nemolizumab previously.
* Participants who are mentally, physically, or linguistically unable to understand the content of the ICF and/or to complete the study questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The clinical decision for treatment with nemolizumab has to be made by the physicians independently of the participation in this NIS and prior to the informed consent process. Participants greater than or equal to (>=) 18 years of age will be eligible for the trial.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Investigator Global Assessment-chronic Prurigo (IGA-CPG stage) at Month 6 | At 6 month
  The IGA-CPG stage is an instrument used to assess the overall number and thickness of chronic prurigo lesions at a given time point, as determined by the physician. In this scale, nodules, papules, plaques, and other PN lesions are defined as pruriginous lesions or chronic prurigo lesions. A single score will be determined by the physician as follows: 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate), or 4 (severe). A higher score indicates severe chronic prurigo.
Peak Pruritus Numerical Rating Scale (PP NRS) at Month 6 | At 6 month
  The PP NRS is a single-question validated PRO assessment that participants will use to report the maximum intensity of their pruritus (itch). The PP NRS consists of the following question: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". Here, a lower score indicates a better outcome.

SECONDARY OUTCOMES:
Investigator Global Assessment-chronic Prurigo (IGA-CPG stage) Up to Month 12 | Up to 12 months
  The IGA-CPG stage is an instrument used to assess the overall number and thickness of chronic prurigo lesions at a given time point, as determined by the physician. In this scale, nodules, papules, plaques, and other PN lesions are defined as pruriginous lesions or chronic prurigo lesions. A single score will be determined by the physician as follows: 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate), or 4 (severe). A higher score indicates severe chronic prurigo.
Prurigo Activity Score (PAS) Up to Month 12 | Up to 12 months
  The PAS is a physician-assessed tool to monitor the distribution and activity of chronic prurigo lesions. This includes a count of the number of lesions in a representative area and a calculated staging (stage 0 to stage 4) based on the percentage of lesions with excoriations/crusts and healed lesions compared to all lesions. A higher score indicates higher level of activity.
Peak Pruritus Numerical Rating Scale (PP NRS) Up to Month 12 | Up to 12 months
  The PP NRS is a single-question validated PRO assessment that participants will use to report the maximum intensity of their pruritus (itch). The PP NRS consists of the following question: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". Here, a lower score indicates a better outcome.
Sleep Disturbance Numerical Rating Scale (SD NRS) Up to Month 12 | Up to 12 months
  The SD NRS is a single-item PRO for quantifying sleep disturbance that has been validated in PN participants. The SD NRS consists of the following question: "On a scale of 0 to 10, with 0 being 'no sleep loss related to the symptoms of my skin disease (prurigo nodularis)' and 10 being 'I did not sleep at all due to the symptoms of my skin disease (prurigo nodularis)', how would you rate your sleep last night". Here, a lower score indicates a better outcome.

CONTACTS AND LOCATIONS:
Locations (51):
- United States (39):
  - Galderma Investigational Site # 8893, Birmingham, Alabama
  - Galderma Investigational Site # 7077, Phoenix, Arizona
  - Galderma Investigational Site # 7060, Phoenix, Arizona
  - Galderma Investigational Site # 7067, Tucson, Arizona
  - Galderma Investigational Site # 7074, Corona, California
  - Galderma Investigational Site # 6836, Fountain Valley, California
  - Galderma Investigational Site # 8224, Fremont, California
  - Galderma Investigational Site # 7064, Santa Monica, California
  - Galderma Investigational Site # 7061, Castle Rock, Colorado
  - Galderma Investigational Site # 7059, Fairfield, Connecticut
  - Galderma Investigational Site # 7087, Coral Gables, Florida
  - Galderma Investigational Site # 7063, Cutler Bay, Florida
  - Galderma Investigational Site # 7078, Miami, Florida
  - Galderma Investigational Site # 7070, North Miami Beach, Florida
  - Galderma Investigational Site # 7091, Tampa, Florida
  - Galderma Investigational Site # 7058, Chicago, Illinois
  - Galderma Investigational Site # 8142, Indianapolis, Indiana
  - Galderma Investigational Site # 8012, Glendale, Maryland
  - Galderma Investigational Site # 7068, Rockville, Maryland
  - Galderma Investigational Site # 7065, Brighton, Massachusetts
  - Galderma Investigational Site # 7066, Auburn Hills, Michigan
  - Galderma Investigational Site # 7071, Caledonia, Michigan
  - Galderma Investigational Site # 7072, Troy, Michigan
  - Galderma Investigational Site # 7053, Waterford, Michigan
  - Galderma Investigational Site # 7057, Lee's Summit, Missouri
  - Galderma Investigational Site # 7076, St Louis, Missouri
  - Galderma Investigational Site # 7055, Portsmouth, New Hampshire
  - Galderma Investigational Site # 7080, Auburn, New York
  - Galderma Investigational Site # 7052, East Syracuse, New York
  - Galderma Investigational Site # 8282, Mount Kisco, New York
  - Galderma Investigational Site # 7056, New York, New York
  - Galderma Investigational Site # 7051, New York, New York
  - Galderma Investigational Site # 7081, Dayton, Ohio
  - Galderma Investigational Site # 8559, Philadelphia, Pennsylvania
  - Galderma Investigational Site # 8238, Dallas, Texas
  - Galderma Investigational Site # 7062, Edinburg, Texas
  - Galderma Investigational Site # 7088, Grapevine, Texas
  - Galderma Investigational Site # 7069, Sugar Land, Texas
  - Galderma Investigational Site # 7079, Vienna, Virginia
- Germany (12):
  - Galderma Investigational Site # 6374, Karlsruhe, Baden-Wurttemberg
  - Galderma Investigational Site # 6369, Erlangen, Bavaria
  - Galderma Investigation Site # 6367, Rostock, Mecklenburg-Vorpommern
  - Galderma Investigational Site # 5437, Kiel, Schleswig-Holstein
  - Galderma Investigational Site # 6387, Ahaus
  - Galderma Investigational Site # 6385, Berlin
  - Galderma Investigational Tracker Site # 6172, Berlin
  - Galderma Investigational Site # 6386, Bielefeld
  - Galderma Investigational Site # 6370, Haslach
  - Galderma Investigational Site # 6384, Koblenz
  - Galderma Investigational Site # 6373, Mainz
  - Galderma Investigational Site # 6371, Oberursel

IPD SHARING:
Plan to Share IPD: Undecided